CLINICAL TRIAL: NCT04212507
Title: The Gut-Skin Axis Integrity in Psoriatic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amal Mohammed Hosni Alameldin Mhmoud, Dr.principal investigator, Assiut University
Other Study IDs: the GSAI in Psoriatic Patients
Record Dates: First submitted 2019-12-24; First posted 2019-12-27 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Psoriatic Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: 50 psoriatic patients
  Interventions: Diagnostic Test: The serum level of Claudin-3 and intestinal Fatty acid binding protein
- 2: 30 age and sex-matched healthy volunteers as a control group
  Interventions: Diagnostic Test: The serum level of Claudin-3 and intestinal Fatty acid binding protein

INTERVENTIONS:
Diagnostic Test: The serum level of Claudin-3 and intestinal Fatty acid binding protein — The serum level of Claudin-3 and intestinal Fatty acid-binding protein between patients with psoriasis and controls Understanding the interplay between microbiota, gut barrier and inflammation may contribute to the development of new methods of preventing onset or exacerbations of psoriasis and new therapeutic approach for psoriasis.
  Other Names: Complete blood count ,Liver enzymes ,Fasting blood glucose and Serum creatinine level

SUMMARY:
Assess two non-invasive markers of intestinal barrier integrity {Claudin-3 and intestinal Fatty acid-binding protein (I-FABP)} in patients with psoriasis and to evaluate the possible relation of these markers with the demographic and clinical data.

DETAILED DESCRIPTION:
Psoriasis is a common non-infectious chronic immune-mediated skin disorder that is associated with the considerable physical and social burden .Its estimated prevalence varies globally and is highest in western countries, where it affects around 2-4% of the population The most common form is plaque psoriasis, accounting 90% of all cases and manifesting as sharply demarcated erythematous plaques covered by silvery scales The gut microbiota refers to the complex community of microorganisms, covering more than 1000 different species of bacteria, viruses, fungi, and protozoa.

The gut commensals predominantly aid in nutrient metabolism, drug metabolism, prevention of colonization of pathogenic microorganisms and in intestinal barrier function..

Dysbiosis or alterations in the composition and function of the microbiota has been implicated in the development and progression of various skin diseases. The concept of "gut-skin axis" links the effects of dysbiosis with many skin diseases.

Disruption of the intestinal barrier can cause translocation of bacteria and their endotoxins or metabolites, which further induces or aggravates systemic inflammation The intestinal barrier function is maintained by a lining of enterocytes and tight junctions, sealing the paracellular space between adjacent enterocytes. Intestinal barrier integrity loss can be assessed by evaluation of intestinal epithelial cell damage or tight junction loss Claudins are transmembrane proteins which participate in the formation of tight junctions by binding to the actin cytoskeleton. Blood Claudin- 3 is considered as a useful early non-invasive biomarker of intestinal permeability due to its small size Fatty acid-binding proteins (FABP) are small (14-15 kDa) cytosolic water-soluble proteins, present in mature enterocytes of the small and large intestine... It is also considered a reliable marker of intestinal barrier integrity Psoriasis is a systemic inflammatory disease with complex multifactorial pathogenesis. Recently, considerable interest has been focused on the interaction between the gut microbiome, intestinal barrier and immune system. The so-called 'gut-skin axis' has been suggested to be a key factor and an interesting area of research in the etiopathogenesis of psoriasis with potential attractive therapeutic implications

ELIGIBILITY:
Inclusion Criteria:

* psoriatic patients and age and sex-matched healthy volunteers as a control group

Exclusion Criteria:

* - History of acute gastrointestinal infection or gastrointestinal surgery during the last 3 months prior to the study
* Intake of probiotics or prebiotics during the last one month.
* Systemic anti-psoriatic treatment in the previous 3 months
* Topical or phototherapy during the last month
* Dietary restrictions during the last 3 months
* Chronic gastrointestinal disorder (celiac disease, inflammatory bowel diseases, irritable bowel disease, food allergies)
* Liver cirrhosis
* Cardiac failure
* Any associated skin or systemic illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: psoriatic patients and age and sex-matched healthy volunteers as a control group
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Compare the serum level of Claudin-3 and intestinal Fatty acid binding protein between patients with psoriasis and controls | Baseline
  Understanding the interplay between microbiota, gut barrier and inflammation to study the aetiopathogenesis of psoriasis may contribute to the development of new methods of preventing onset or exacerbations of psoriasis and new therapeutic approach for psoriasis.

REFERENCES:
- [Background] Traks T, Keermann M, Prans E, Karelson M, Loite U, Koks G, Silm H, Koks S, Kingo K. Polymorphisms in IL36G gene are associated with plaque psoriasis. BMC Med Genet. 2019 Jan 11;20(1):10. doi: 10.1186/s12881-018-0742-2. PMID 30634937
- [Background] Jandhyala SM, Talukdar R, Subramanyam C, Vuyyuru H, Sasikala M, Nageshwar Reddy D. Role of the normal gut microbiota. World J Gastroenterol. 2015 Aug 7;21(29):8787-803. doi: 10.3748/wjg.v21.i29.8787. PMID 26269668
- [Background] Barmeyer C, Fromm M, Schulzke JD. Active and passive involvement of claudins in the pathophysiology of intestinal inflammatory diseases. Pflugers Arch. 2017 Jan;469(1):15-26. doi: 10.1007/s00424-016-1914-6. Epub 2016 Nov 30. PMID 27904960
- [Background] Salem I, Ramser A, Isham N, Ghannoum MA. The Gut Microbiome as a Major Regulator of the Gut-Skin Axis. Front Microbiol. 2018 Jul 10;9:1459. doi: 10.3389/fmicb.2018.01459. eCollection 2018. PMID 30042740